CLINICAL TRIAL: NCT05965856
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B003 Monotherapy and BL-B01D1+SI-B003 Combination Therapy (BL-B01D1+SI-B003) in Patients With Locally Advanced or Metastatic Urothelial Carcinoma and Other Solid Tumors
Brief Title: A Study of SI-B003 and BL-B01D1+SI-B003 in Patients With Locally Advanced or Metastatic Urothelial Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-06
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Urothelial Carcinoma; Solid Tumor
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 + SI-B003 (Experimental): Participants receive SI-B003 or BL-B01D1+SI-B003 dual therapy in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — Administration by intravenous infusion

SUMMARY:
This phase II study is designed to explore the efficacy and safety of SI-B003 monotherapy and BL-B01D1+SI-B003 combination therapy in patients with locally advanced or metastatic urothelial carcinoma and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects voluntarily participated in the study and signed informed consent;
2. Male or female aged ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG 0-1;
5. Locally advanced or metastatic urothelial carcinoma and other solid tumors confirmed by histopathology and/or cytology who have failed or cannot tolerate standard treatment or who currently have no standard treatment or cannot obtain standard treatment; (including but not limited to urothelial cancer, prostate cancer, kidney cancer) : ① Urothelial cancer should have received previous failure or intolerance to standard platinum-based chemotherapy; ② Prostate cancer with pathological type of adenocarcinoma should have received at least one previous novel hormonal therapy (abiraterone acetate, enzalutamide, etc.) and at least one failed or intolerant taxane regimen (docetaxel, cabazitaxel); ③ Clear cell renal cell carcinoma required previous failure or intolerance to standard first-line tyrosine kinase inhibitor (TKI) regimens. ④ Locally advanced or metastatic other urological malignancies (non-clear cell renal cancer, penile cancer, etc.) that failed standard treatment and were not suitable for surgery or radiotherapy. Treatment failure was defined as disease progression during or after treatment with systemic antitumor regimens. Intolerance refers to patients who have received standard treatment and have grade 3-4 adverse reactions, and refuse to continue the original regimen.

   Note: Recurrence or disease progression within 6 months of the last chemotherapy in multimodal therapy was considered as first-line treatment.
6. Consent to provide archival tumor tissue specimens (10 unstained sections (anti-slip) surgical specimens (thickness 4-5μm)) or fresh tissue samples from primary or metastatic lesions within 3 years. If participants cannot provide tumor tissue samples, they can be enrolled if they meet other inclusion and exclusion criteria, after the evaluation of the investigator;
7. Must have at least one measurable lesion according to RECIST v1.1 definition; Lesions that had been previously treated with radiation could be included in a measurable lesion only if there was definite disease progression after radiation therapy.
8. Provided that no blood transfusions and no use of any cell growth factors and/or platelet-raising agents are allowed for 14 days prior to the screening period, organ function levels must meet the following criteria:

   1. Blood routine: hemoglobin (HGB) ≥ 90g/L; Absolute neutrophil count (NEUT) ≥1.5×10 9 /L; Platelet count (PLT) ≥ 100×10 9 /L;
   2. Renal function: creatinine (Cr) ≤1.5 ULN, or creatinine clearance (Ccr) ≥40 mL/min (according to Cockcroft and Gault formula).
   3. Liver function: total bilirubin (TBIL≤1.5 ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) were all ≤2.5 ULN, and AST and ALT were both ≤5.0 ULN when liver metastasis was present;
   4. Coagulation function: international normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5ULN;
   5. no severe cardiac dysfunction with left ventricular ejection fraction ≥50%;
9. Toxicity from previous antineoplastic therapy has returned to grade 1 or less as defined by NCI-CTCAE v5.0 (asymptomatic laboratory abnormalities such as ALP elevation, hyperuricemia, and hyperglycemia were considered by the investigator, and toxicity with no safety risk was judged by the investigator; Except for alopecia, grade 2 peripheral neurotoxicity, or decreased hemoglobin ≥90g/L).
10. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before the start of treatment, the serum or urine pregnancy test must be negative, and the patient must not be lactating; All enrolled patients should take adequate barrier contraception during the entire treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Previous use of an ADC drug with a topoisomerase I inhibitor as a toxin;
2. Administration of chemotherapy or chemotherapy within 4 weeks or 5 half-lives, whichever is shorter, before the first dose Physical therapy, immunotherapy, definitive radiotherapy, major surgery (investigator's definition), targeted therapy (including Small molecule tyrosine kinase inhibitors) and other anti-tumor therapy; Mitomycin and nitrosoureas were given for the first time Within 6 weeks before treatment; Oral fluorouracil drugs such as S-1, capecitabine, or palliative radiotherapy for Within 2 weeks before the first dose; No exposure to wide-field radiotherapy within 4 weeks before study treatment for prostate cancer (tired) And ≥30% bone marrow), samarium must be completed 4 weeks prior to the first dose of treatment, and strontium and Lu 177 treatment This must be completed at least 12 weeks before the first administration of treatment, and radium-233 must precede the first administration of treatment At least 6 weeks to complete. Prostate cancer bone metastasis therapy such as bisphosphonates or denosumab should be administered before the first dose It was initiated at 4 weeks and was administered at a stable dose.
3. Patients with a history of immunotherapy and grade ≥3 irAE or grade ≥2 immune-related myocarditis must be excluded;
4. Use of immunomodulatory drugs within 14 days before the first use of the study drug, including but not limited to thymosin, Interleukin-2, interferon, etc. must be excluded;
5. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias or grade III atria requiring clinical intervention Ventricular block;
   2. prolonged QT interval at rest (QTc > 450 msec in men or QTc > 470 msec in women);
   3. cerebrovascular accident or transient ischemic attack within 6 months before the first dose; Symptomatic congestive History of heart failure (CHF) ≥ grade 2 (CTCAE 5.0) and New York Heart Association (NYHA) ≥ Grade 2 heart failure, transmural myocardial infarction history, unstable angina, etc.
6. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, requiring systemic treatment Psoriasis, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, etc., excluding type I sugar Urinary disorders, hypothyroidism that can be controlled with replacement therapy alone, skin disorders that do not require systemic treatment (e.g Vitiligo and psoriasis).
7. Systemic corticosteroids (> 10mg/ day prednisone, or equivalent) are required within 2 weeks before the study dose Doses of other corticosteroids) or immunosuppressive agents; Inhaled or topical administration of hormones, or due to adrenal The exception is those who were treated with physiological replacement doses of hormone for insufficiency;
8. Other malignancies that progressed or required treatment within 5 years before the first dose, such as the following External: radical resection of skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, radical resection of carcinoma in situ, such as breast carcinoma in situ, prostate cancer; Remarks: Localized low-risk prostate cancer (Defined as stage ≤T2a, Gleason score ≤6, and PSA < 10ng/mL at prostate cancer diagnosis (e.g Measured) had received curative treatment and had no PSA biochemical recurrence Were eligible to participate in this study);
9. History of (noninfectious) interstitial lung disease (ILD)/pulmonary inflammation requiring steroid therapy, or when Patients with previous ILD/ pulmonary inflammation, or suspected ILD/ pulmonary inflammation that could not be excluded by imaging at the time of screening Syndrome;
10. Prior to starting the study treatment, there are:

    1. Poorly controlled diabetes (fasting blood glucose ≥ 13.3 mmol/L)
    2. Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
    3. History of hypertensive crisis or hypertensive encephalopathy
11. Unstable deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening Thrombotic events such as plug; Infusion-related thrombosis was excluded.
12. Patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases). But he had a brain turn Metastatic therapy (radiotherapy or surgery; And the subjects had stopped radiotherapy and surgery 2 weeks before the first dose.) Patients with stable brain metastases less than 10mm in diameter were eligible for enrollment Patients (with leptomeningeal metastases) were excluded even if they were treated and judged to be stable.
13. Patients with large amount of serous cavity effusion, or serous cavity effusion with symptoms, or before signing informed consent Patients who underwent drainage within 4 weeks;
14. Allergic history to recombinant humanized antibody or human-mouse chimeric antibody or to BL-B01D1, SI-B003 Patients who are allergic to excipients;
15. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus Infection (HBV-DNA copy number > 103 IU/ml) or active hepatitis C virus infection (anti-HCV Body positive and HCV-RNA > detection limit).
17. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.
18. Participated in another clinical trial within 4 weeks before the first dose (calculated from the time of the last dose);
19. Persons who have a history of psychotropic drug abuse and cannot be abstinent or have mental disorders;
20. Any other circumstances that the investigator deemed inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B003.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China